CLINICAL TRIAL: NCT04124042
Title: A Double-Blind, Placebo-Controlled Assessment of the Tolerability and Efficacy of XT-150 for the Treatment of Moderate to Severe Pain Due to Osteoarthritis of the Knee
Brief Title: Efficacy and Safety of XT-150 in Osteoarthritis of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xalud Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XT-150-2-0204
Record Dates: First submitted 2019-10-09; First posted 2019-10-11 (Actual); Results first posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-01

CONDITIONS: Osteoarthritis, Knee
Keywords: Inflammation; Pain; Interleukin; Gene Therapy; plasmid DNA
MeSH Terms: conditions — Osteoarthritis, Knee; Inflammation; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Stage A: 0.15 mg/mL XT-150, Stage B: 0.15 mg/mL XT-150 (Experimental): Low dose active in Stage A and Stage B
  Interventions: Biological: XT-150
- Stage A: 0.15 mg/mL XT-150, Stage B: 0.45 mg/mL XT-150 (Experimental): Low dose active in Stage A, high dose active in Stage B
  Interventions: Biological: XT-150
- Stage A: 0.45 mg/mL XT-150, Stage B: 0.15 mg/mL XT-150 (Experimental): High dose active in Stage A, low dose active in Stage B
  Interventions: Biological: XT-150
- Stage A: 0.45 mg/mL XT-150, Stage B: 0.45 mg/mL XT-150 (Experimental): High dose active in Stage A and Stage B
  Interventions: Biological: XT-150
- Stage A: Placebo, Stage B: 0.15 mg/mL XT-150 (Placebo Comparator): Inactive comparator in Stage A, low dose active in Stage B
  Interventions: Biological: XT-150; Drug: Placebo
- Stage A: Placebo, Stage B: 0.45 mg/mL XT-150 (Placebo Comparator): Inactive comparator in Stage A, high dose active in Stage B
  Interventions: Biological: XT-150; Drug: Placebo

INTERVENTIONS:
Biological: XT-150 — plasmid DNA
Drug: Placebo — Placebo is a sterile phosphate-buffered saline
  Arms: Stage A: Placebo, Stage B: 0.15 mg/mL XT-150; Stage A: Placebo, Stage B: 0.45 mg/mL XT-150

SUMMARY:
This is a Phase 2 safety and efficacy study of XT-150 in adult participants experiencing moderate to severe pain due to osteoarthritis of the knee.

DETAILED DESCRIPTION:
In this Phase 2 study, Baseline (Day 0) confirmation of study eligibility will be completed the day before or day of study drug administration.

Study drug will be administered by intra-articular (IA) injection into the joint space of the index knee (knee selected for treatment).

Up to 270 participants will be randomly enrolled into 1 of 6 treatment sequences (45 participants/ group). Treatment Groups:

1. 0.15 mg/mL XT-150 (1mL), 0.15 mg/mL XT-150 (1mL)
2. 0.15 mg/mL XT-150 (1mL), 0.45 mg/mL XT-150 (1mL)
3. 0.45 mg/mL XT-150 (1mL), 0.15 mg/mL XT-150 (1mL)
4. 0.45 mg/mL XT-150 (1mL), 0.45 mg/mL XT-150 (1mL)
5. Placebo (1mL), 0.15 mg/mL XT-150 (1mL)
6. Placebo (1mL), 0.45 mg/mL XT-150 (1mL)

The study will be conducted in 2 stages, A and B. Participants will be randomized at Day 0 to a treatment regimen, one treatment assignment for Stage A and one treatment assignment for Stage B:

Stage A (Up to Day 180): Participants will receive placebo, 0.15 mg/mL XT-150 or 0.45 mg/mL XT-150 to the index knee at Day 0.

Stage B (Day 180 to Day 360): Participants will have the option to receive a pre-randomized dose (XT-150 0.15 mg/mL or 0.45 mg/mL) to the index knee anytime between Day 180 and Day 330.

Final assessments will be 12 months after the first IA dose.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic disease due to osteoarthritis, defined as a WOMAC Pain score ≥ 8 (worst possible = 20)
2. Focused Analgesia Selection Test will be used to determine whether patients can report pain with sufficient consistency to enter the clinical trial
3. Males and females between 45 and 85 years of age, inclusive
4. Kellgren-Lawrence grading of 2 or 3 within the last 6 months
5. Stable analgesic regimen during the 4 weeks prior to enrollment
6. In the judgment of the Investigator, acceptable general medical condition
7. Life expectancy >6 months
8. Male and female participants who are heterosexually active and not surgically sterile must agree to use effective contraception, including abstinence, for the duration of the study
9. Have suitable knee joint anatomy for intra-articular injection
10. Willing and able to return for the follow-up (FU) visits
11. Able to read and understand study instructions, and willing and able to comply with all study procedures

Exclusion Criteria:

1. Hypersensitivity, allergy, or significant reaction to any ingredient of the study drug, including double-stranded DNA, mannose, and sucrose
2. Previously received XT-150 injection(s)
3. Scheduled partial or complete knee replacement within 6 months; participant agrees not to schedule a knee replacement during Stage A of the study
4. History of knee arthroplasty on the Index Knee, i.e., selected for study injection(s)
5. History of rheumatoid arthritis or other inflammatory disease
6. History of immunosuppressive therapy; systemic steroids in the last 3 months
7. Received knee injection with hyaluronic acid or stem-cells in the last 6 months
8. Knee injection of glucocorticoid in the last 3 months
9. Current treatment with systemic immunosuppressive (systemic corticosteroid therapy or other strong immunosuppressant)
10. Currently receiving systemic chemotherapy or radiation therapy for malignancy
11. Clinically significant hepatic disease as indicated by clinical laboratory results ≥3 times the upper limit of normal for any liver function test (e.g., aspartate aminotransferase, alanine aminotransferase)
12. Severe anemia (Grade 3; hemoglobin <8.0 g/dL, <4.9 mmol/L, <80 g/L; transfusion indicated), Grade 1 white cell counts (lymphocytes <LLN - 800/mm^3; <LLN - 0.8 x 109 /L, neutrophils <LLN - 1500/mm^3; <LLN - 1.5 x 109 /L), LLN=Lower Limit Normal Range
13. Positive serology for human immunodeficiency virus, hepatitis B virus, or hepatitis C virus
14. Significant neuropsychiatric conditions; dementia, major depression, or altered mental state that in the opinion of the Investigator will interfere with study participation
15. Current treatment with systemic antibiotics or antivirals (EXCEPTION: topical treatments)
16. Current anticoagulant or anti-platelet treatment (e.g., warfarin, heparins, factor X inhibitors, clopidogrel, prasugrel, ticagrelor, or dipyridamole). Low-dose (≤ 325 mg/day) aspirin is permitted
17. Known or suspected history of active alcohol or intravenous/oral drug abuse within 1 year before the screening visit
18. Use of any investigational drug or device within 3 months before enrollment or current participation in a trial that included intervention with a drug or device; or currently participating in an investigational drug or device study
19. Any condition that, in the opinion of the Investigator, could compromise the safety of the participant, the participant's ability to communicate with the study staff, or the quality of the data

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-04-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (4):
  - eStudySite, La Mesa, California
  - Neurovations (Napa Pain Institute), Napa, California
  - Source Healthcare, Santa Monica, California
  - Carolinas Clinical Research Institute, Winston-Salem, North Carolina
- Australia (2):
  - University of Adelaide in collaboration with CMAX Clinical Research Pty Ltd, Adelaide, South Australia
  - Alfred Health, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen L, Huang FL, Tang Q, Zhao ZK, Ye ZY, Liang JH. Targeted therapy for knee osteoarthritis: From basic to clinics. Medicine (Baltimore). 2025 Aug 15;104(33):e43686. doi: 10.1097/MD.0000000000043686. PMID 40826764

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 289 participants signed a consent form, but 3 withdrew during the screening period. 286 participants were dosed and that is the number reflected in this section. The data listed here is based on the Safety Population and actual treatment received, not the ITT population. One participant received 0.15mg due to a site error, although they were originally randomized to 0.45mg in Stage A.
Period: Overall Study
Arm/Group | Stage A: 0.15 mg/mL XT-150, Stage B: 0.15 mg/mL XT-150 | Stage A: 0.15 mg/mL XT-150, Stage B: 0.45 mg/mL XT-150 | Stage A: 0.45 mg/mL XT-150, Stage B: 0.15 mg/mL XT-150 | Stage A: 0.45 mg/mL XT-150, Stage B: 0.45 mg/mL XT-150 | Stage A: Placebo, Stage B: 0.15 mg/mL XT-150 | Stage A: Placebo, Stage B: 0.45 mg/mL XT-150
Started (The number of participants listed here is based on the Safety Population and actual treatment received, not the ITT population. One participant received 0.15mg due to a site error, although they were originally randomized to 0.45mg in Stage A.) | 49 | 47 | 47 | 47 | 48 | 48
Completed | 39 | 42 | 38 | 39 | 42 | 43
Not Completed | 10 | 5 | 9 | 8 | 6 | 5

BASELINE CHARACTERISTICS:
Population: The number of participants listed here is based on the Safety Population and actual treatment received, not the ITT population. One participant received 0.15mg due to a site error, although they were originally randomized to 0.45mg in Stage A.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage A: 0.15 mg/mL XT-150, Stage B: 0.15 mg/mL XT-150 | Stage A: 0.15 mg/mL XT-150, Stage B: 0.45 mg/mL XT-150 | Stage A: 0.45 mg/mL XT-150, Stage B: 0.15 mg/mL XT-150 | Stage A: 0.45 mg/mL XT-150, Stage B: 0.45 mg/mL XT-150 | Stage A: Placebo, Stage B: 0.15 mg/mL XT-150 | Stage A: Placebo, Stage B: 0.45 mg/mL XT-150 | Total
Number analyzed (Participants) | 49 | 47 | 47 | 47 | 48 | 48 | 286
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (8.15) | 62.0 (6.68) | 64.9 (7.09) | 62.6 (7.82) | 62.9 (7.35) | 65.3 (9.52) | 63.3 (7.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 22 | 33 | 27 | 33 | 155
  Male | 29 | 27 | 25 | 14 | 21 | 15 | 131
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 0 | 0 | 1 | 2 | 14
  Not Hispanic or Latino | 42 | 43 | 47 | 47 | 47 | 46 | 272
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 1 | 2 | 0 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 10 | 6 | 5 | 5 | 11 | 4 | 41
  White | 35 | 41 | 39 | 38 | 31 | 39 | 223
  More than one race | 3 | 0 | 2 | 2 | 3 | 2 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 2 | 0 | 2
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 32.482 (7.398) | 31.823 (7.087) | 31.101 (7.192) | 33.401 (8.190) | 32.405 (5.234) | 31.659 (7.236) | 32.150 (7.047)

OUTCOME MEASURES:

1. Primary Outcome: Stage A: Number of Participants Achieving 30% Improvement From Baseline in Western Ontario and McMasters Arthritis Index (WOMAC) Pain Score
Description: The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score will be obtained from the Knee injury and Osteoarthritis Outcome Score (KOOS) questionnaire which is a validated, commonly used instrument to assess the participant's opinion about their knee and associated problems. Each item is answered on a 5-point Likert scale. The score for pain category ranges from 0 (no pain) to 20 (maximum pain); higher score indicates worse outcomes. Baseline is defined as the Day 0 value.
Time Frame: Day 180
Population: The Intent-to-Treat (ITT) Population will comprise all enrolled participants who received the treatment injection, analyzed according to randomized Stage A treatment. The ITT Population will be the primary analysis population for efficacy.
  One (1) participant was randomized to 0.45 mg/ml XT-150 but inadvertently received 0.15 mg/ml XT-150 due to site error, explaining the difference between number analyzed in XT-150 groups compared to the overall participant flow.
Measure: Count of Participants; unit: Participants
Groups:
- Stage A: 0.15 mg/ml XT-150: Low dose active in Stage A
- Stage A: 0.45 mg/ml XT-150: High dose active in Stage A
- Stage A: Placebo: Inactive comparator in Stage A
Arm/Group | Stage A: 0.15 mg/ml XT-150 | Stage A: 0.45 mg/ml XT-150 | Stage A: Placebo
Number analyzed (Participants) | 95 | 95 | 96
Participants
  Responder | 26 | 28 | 38
  Non-responder | 53 | 56 | 51
  Not Analyzed | 16 | 11 | 7
Statistical Analysis 1: Comparison: Stage A: 0.15 mg/ml XT-150 vs Stage A: Placebo; Test type: Superiority; Odds Ratio (OR) = 0.655, 95% CI 2-sided [0.347 to 1.237]
Statistical Analysis 2: Comparison: Stage A: 0.45 mg/ml XT-150 vs Stage A: Placebo; Test type: Superiority; Odds Ratio (OR) = 0.714, 95% CI 2-sided [0.381 to 1.336]

2. Primary Outcome: Stage A: Change From Baseline in WOMAC Pain Score at Day 180
Description: as for outcome 1
Time Frame: Day 180
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Stage A: 0.15 mg/ml XT-150 | Stage A: 0.45 mg/ml XT-150 | Stage A: Placebo
Number analyzed (Participants) | 95 | 95 | 96
score on a scale | -1.77 (0.386) | -1.95 (0.380) | -2.21 (0.374)
Statistical Analysis 1: Comparison: Stage A: 0.15 mg/ml XT-150 vs Stage A: Placebo; Test type: Superiority; p = 0.413, Mixed Models Analysis; Mean Difference (Final Values) = 0.44, 95% CI 2-sided [-0.62 to 1.50], Standard Error of Mean 0.539
Statistical Analysis 2: Comparison: Stage A: 0.45 mg/ml XT-150 vs Stage A: Placebo; Test type: Superiority; p = 0.629, Mixed Models Analysis; Mean Difference (Final Values) = 0.26, 95% CI 2-sided [-0.79 to 1.31], Standard Error of Mean 0.535

3. Primary Outcome: Stage A: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Adverse events were collected from the time of informed consent through the last study visit on Day 360 (1 year). Treatment Emergent Adverse Events (TEAEs) occurred from the time of study drug treatment on Day 0 through end of study (Day 360) or early termination. This analysis reports any AEs/SAEs that occurred prior to the second dose.
Time Frame: Prior to second dose (Up to Day 180-Day 330)
Population: The Safety Population will comprise all participants who receive any amount of study drug, analyzed according to treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage A: 0.15 mg/ml XT-150 | Stage A: 0.45 mg/ml XT-150 | Stage A: Placebo
Number analyzed (Participants) | 96 | 94 | 96
Participants
  Any TEAEs: Yes | 30 | 53 | 38
  Any TEAEs: No | 66 | 41 | 58
  Related TEAEs: Yes | 4 | 0 | 4
  Related TEAEs: No | 92 | 94 | 92
  Serious TEAEs: Yes | 2 | 3 | 6
  Serious TEAEs: No | 94 | 91 | 90
  Related Serious TEAEs: Yes | 0 | 0 | 0
  Related Serious TEAEs: No | 96 | 94 | 96

4. Primary Outcome: Stage B: Number of Participants With AEs and SAEs
Description: Adverse events were collected from the time of informed consent through the last study visit on Day 360 (1 year). Treatment Emergent Adverse Events occurred from the time of study drug treatment on Day 0 through end of study (Day 360) or early termination. This analysis reports any AEs/SAEs that occurred after the second dose.
Time Frame: Post Second Dose (Day 180-Day 330 through Day 360)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Stage A: 0.15 mg/mL XT-150, Stage B: 0.15 mg/mL XT-150 | Stage A: 0.15 mg/mL XT-150, Stage B: 0.45 mg/mL XT-150 | Stage A: 0.45 mg/mL XT-150, Stage B: 0.15 mg/mL XT-150 | Stage A: 0.45 mg/mL XT-150, Stage B: 0.45 mg/mL XT-150 | Stage A: Placebo, Stage B: 0.15 mg/mL XT-150 | Stage A: Placebo, Stage B: 0.45 mg/mL XT-150
Number analyzed (Participants) | 39 | 41 | 37 | 41 | 43 | 43
Participants
  Any TEAE: Yes | 12 | 14 | 18 | 16 | 9 | 18
  Any TEAE: No | 27 | 27 | 19 | 25 | 34 | 25
  Related TEAE: Yes | 0 | 0 | 0 | 1 | 0 | 1
  Related TEAE: No | 39 | 41 | 37 | 40 | 43 | 42
  Serious TEAE: Yes | 2 | 1 | 1 | 1 | 0 | 1
  Serious TEAE: No | 37 | 40 | 36 | 40 | 43 | 42
  Related Serious TEAE: Yes | 0 | 0 | 0 | 0 | 0 | 0
  Related Serious TEAE: No | 39 | 41 | 37 | 41 | 43 | 43

5. Secondary Outcome: Stage B: Change From Baseline in WOMAC Pain Score at Day 360
Description: as for outcome 1
Time Frame: Day 360
Population: The Intent-to-Treat (ITT) Population will comprise all enrolled participants who received the treatment injection, analyzed according to randomized Stage A treatment. The ITT Population will be the primary analysis population for efficacy.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Stage A: 0.15 mg/mL XT-150, Stage B: 0.15 mg/mL XT-150 | Stage A: 0.15 mg/mL XT-150, Stage B: 0.45 mg/mL XT-150 | Stage A: 0.45 mg/mL XT-150, Stage B: 0.15 mg/mL XT-150 | Stage A: 0.45 mg/mL XT-150, Stage B: 0.45 mg/mL XT-150 | Stage A: Placebo, Stage B: 0.15 mg/mL XT-150 | Stage A: Placebo, Stage B: 0.45 mg/mL XT-150
Number analyzed (Participants) | 39 | 41 | 38 | 40 | 42 | 43
score on a scale | -3.4 (0.666) | -3.26 (0.662) | -3.44 (0.682) | -3.87 (0.643) | -2.9 (0.659) | -2.9 (0.639)

6. Secondary Outcome: Stage B: Change From Baseline in WOMAC Function Score
Description: The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) function score will be obtained from the Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire which is a is a validated, commonly used instrument to assess the participant's opinion about their knee and associated problems. Each item is answered on a 5-point Likert scale. The function dimension category asks about the degree of difficulty in doing 17 activities. The score ranges from 0 (normal function) to 170 (severely limited function); higher score indicates worse outcomes. Baseline is defined as the Day 0 value.
Time Frame: At Day 360
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Stage A: 0.15 mg/mL XT-150, Stage B: 0.15 mg/mL XT-150 | Stage A: 0.15 mg/mL XT-150, Stage B: 0.45 mg/mL XT-150 | Stage A: 0.45 mg/mL XT-150, Stage B: 0.15 mg/mL XT-150 | Stage A: 0.45 mg/mL XT-150, Stage B: 0.45 mg/mL XT-150 | Stage A: Placebo, Stage B: 0.15 mg/mL XT-150 | Stage A: Placebo, Stage B: 0.45 mg/mL XT-150
Number analyzed (Participants) | 38 | 40 | 36 | 38 | 40 | 43
score on a scale | -11.23 (2.236) | -11.79 (2.292) | -12.8 (2.330) | -13.63 (2.218) | -9.44 (2.292) | -8.66 (2.164)

7. Secondary Outcome: Stage A: Change From Baseline in Brief Pain Inventory (BPI) of Interference Score
Description: The Brief Pain Inventory (BPI) is a self-administered questionnaire for participants to rate the degree to which their pain interferes with common dimensions of feeling and function. The 7 pain interference items will be rated on 0-10 scale. Total interference score ranges from 0 (does not interfere) to 10 (completely interferes); higher score indicates worse outcomes.
Time Frame: Day 180
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Stage A: 0.15 mg/ml XT-150 | Stage A: 0.45 mg/ml XT-150 | Stage A: Placebo
Number analyzed (Participants) | 95 | 95 | 96
score on a scale | -0.96 (0.263) | -1.10 (0.253) | -1.46 (0.258)
Statistical Analysis 1: Comparison: Stage A: 0.15 mg/ml XT-150 vs Stage A: Placebo; Test type: Superiority; p = 0.1374, Mixed Models Analysis; Mean Difference (Final Values) = 0.50, 95% CI 2-sided [-0.16 to 1.16]
Statistical Analysis 2: Comparison: Stage A: 0.45 mg/ml XT-150 vs Stage A: Placebo; Test type: Superiority; p = 0.2807, Mixed Models Analysis; Mean Difference (Final Values) = 0.35, 95% CI 2-sided [-0.29 to 1.00]

8. Secondary Outcome: Stage A: Change From Baseline in Patients Overall Assessment (POA)
Description: The Patient Overall Assessment (POA) is a self-administered questionnaire that records participants' responses to the question "Considering all the ways the OA in your knee affects you, how are you doing today?" on a scale of 1 to 5; 1 being very good (asymptomatic and no limitation of normal activities) to 5, very poor (very severe, intolerable symptoms and inability to carry out normal activities). Higher score indicates worse symptoms.
Time Frame: Day 180
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Stage A: 0.15 mg/ml XT-150 | Stage A: 0.45 mg/ml XT-150 | Stage A: Placebo
Number analyzed (Participants) | 95 | 95 | 96
score on a scale | -0.19 (0.102) | -0.32 (0.100) | -0.33 (0.098)
Statistical Analysis 1: Comparison: Stage A: 0.15 mg/ml XT-150 vs Stage A: Placebo; Test type: Superiority; p = 0.346, Mixed Models Analysis; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.14 to 0.41], Standard Error of Mean 0.142
Statistical Analysis 2: Comparison: Stage A: 0.45 mg/ml XT-150 vs Stage A: Placebo; Test type: Superiority; p = 0.968, Mixed Models Analysis; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.27 to 0.28], Standard Error of Mean 0.140

9. Secondary Outcome: Stage A and B: Number of Participants With Presence of Anti-interleukin (IL)-10 Antibody
Description: Presence of Immunoglobulin M (IgM) or Immunoglobulin G (IgG) antibodies against human IL-10 in serum was assessed at Baseline/Day 0 and then post-initial dose on Days 7, 30, 60, 180, and 360.
Time Frame: Up to Day 360
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Stage A: 0.15 mg/mL XT-150, Stage B: 0.15 mg/mL XT-150 | Stage A: 0.15 mg/mL XT-150, Stage B: 0.45 mg/mL XT-150 | Stage A: 0.45 mg/mL XT-150, Stage B: 0.15 mg/mL XT-150 | Stage A: 0.45 mg/mL XT-150, Stage B: 0.45 mg/mL XT-150 | Stage A: Placebo, Stage B: 0.15 mg/mL XT-150 | Stage A: Placebo, Stage B: 0.45 mg/mL XT-150
Number analyzed (Participants) | 49 | 47 | 47 | 47 | 48 | 48
Participants
  Anti-IL-10 Antibodies Detected | 0 | 0 | 0 | 0 | 0 | 0
  No Anti-IL-10 Antibodies Detected | 49 | 47 | 47 | 47 | 48 | 48

10. Post Hoc Outcome: Post-Hoc WOMAC Pain Score Change From Baseline - 2-dose 0.45mg XT-150 vs. Single-dose 0.45mg XT-150 (mITT)
Description: The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score will be obtained from the Knee injury and Osteoarthritis Outcome Score (KOOS) questionnaire which is a validated, commonly used instrument to assess the participant's opinion about their knee and associated problems. Each item is answered on a 5-point Likert scale. The score for pain category ranges from 0 (no pain) to 20 (maximum pain); higher score indicates worse outcomes. Baseline is defined as the Day 0 value.
  The data reported in this outcome measure is a head-to-head comparison of two doses of 0.45 mg/ml vs. a single dose of 0.45 mg/ml and only includes these 2 treatment sequences whereas outcome measure #12 reports the least squared mean based on data for all 6 treatment sequences.
Time Frame: Day 360
Population: The Modified Intent-to-Treat population consists of the ITT population who received at least one treatment injection with a baseline WOMAC Pain score of 9-20 (>8). This is the target population of interest who may benefit most from the treatment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Stage A: 0.45 mg/mL XT-150, Stage B: 0.45 mg/mL XT-150 | Stage A: Placebo, Stage B: 0.45 mg/mL XT-150
Number analyzed (Participants) | 36 | 29
score on a scale | -5.02 (0.815) | -2.19 (0.911)
Statistical Analysis 1: Comparison: Stage A: 0.45 mg/mL XT-150, Stage B: 0.45 mg/mL XT-150 vs Stage A: Placebo, Stage B: 0.45 mg/mL XT-150; Outcome measure #10 is an analysis of 2 tx groups (two doses of 0.45 mg/ml vs. a single dose of 0.45 mg/ml), whereas outcome measure #12 is all 6 tx groups. A MMRM model was used. LS Means in an MMRM model are influenced by the overall mean structure and covariance estimation. When fewer treatment groups are included, the model adjusts based on a different subset of data, leading to potential shifts in estimated LS Means due to changes in the reference population/covariance structure; Test type: Superiority; p = 0.0081, Mixed Models Analysis; Mean Difference (Final Values) = -2.83, 95% CI 2-sided [-4.91 to -0.75]

11. Post Hoc Outcome: Post-Hoc WOMAC Function Score Change From Baseline - 2-dose 0.45mg XT-150 vs. Single-dose 0.45mg XT-150 (mITT)
Description: The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) function score will be obtained from the Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire which is a is a validated, commonly used instrument to assess the participant's opinion about their knee and associated problems. Each item is answered on a 5-point Likert scale. The function dimension category asks about the degree of difficulty in doing 17 activities. The score ranges from 0 (normal function) to 170 (severely limited function); higher score indicates worse outcomes. Baseline is defined as the Day 0 value.
  The data reported in this outcome measure is a head-to-head comparison of two doses of 0.45 mg/ml vs. a single dose of 0.45 mg/ml and only includes these 2 treatment sequences whereas outcome measure #13 reports the least squared mean based on data for all 6 treatment sequences.
Time Frame: Day 360
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Stage A: 0.45 mg/mL XT-150, Stage B: 0.45 mg/mL XT-150 | Stage A: Placebo, Stage B: 0.45 mg/mL XT-150
Number analyzed (Participants) | 36 | 29
score on a scale | -15.42 (2.887) | -5.82 (3.201)
Statistical Analysis 1: Comparison: Stage A: 0.45 mg/mL XT-150, Stage B: 0.45 mg/mL XT-150 vs Stage A: Placebo, Stage B: 0.45 mg/mL XT-150; Outcome measure #11 is an analysis of 2 tx groups (two doses of 0.45 mg/ml vs. a single dose of 0.45 mg/ml), whereas outcome measure #13 is all 6 tx groups. A MMRM model was used. LS Means in an MMRM model are influenced by the overall mean structure and covariance estimation. When fewer treatment groups are included, the model adjusts based on a different subset of data, leading to potential shifts in estimated LS Means due to changes in the reference population/covariance structure; Test type: Superiority; p = 0.0101, Mixed Models Analysis; Mean Difference (Final Values) = -9.60, 95% CI 2-sided [-16.85 to -2.34]

12. Post Hoc Outcome: Post-Hoc WOMAC Pain Score Change From Baseline - All Dose Regimens (mITT)
Description: as for outcome 1
Time Frame: Day 360
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Stage A: 0.15 mg/mL XT-150, Stage B: 0.15 mg/mL XT-150 | Stage A: 0.15 mg/mL XT-150, Stage B: 0.45 mg/mL XT-150 | Stage A: 0.45 mg/mL XT-150, Stage B: 0.15 mg/mL XT-150 | Stage A: 0.45 mg/mL XT-150, Stage B: 0.45 mg/mL XT-150 | Stage A: Placebo, Stage B: 0.15 mg/mL XT-150 | Stage A: Placebo, Stage B: 0.45 mg/mL XT-150
Number analyzed (Participants) | 35 | 35 | 39 | 36 | 36 | 29
score on a scale | -3.76 (0.835) | -3.53 (0.800) | -4.07 (0.797) | -4.93 (0.789) | -3.03 (0.805) | -2.42 (0.852)

13. Post Hoc Outcome: Post-Hoc WOMAC Function Score Change From Baseline - All Dose Regimens (mITT)
Description: as for outcome 6
Time Frame: Day 360
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Stage A: 0.15 mg/mL XT-150, Stage B: 0.15 mg/mL XT-150 | Stage A: 0.15 mg/mL XT-150, Stage B: 0.45 mg/mL XT-150 | Stage A: 0.45 mg/mL XT-150, Stage B: 0.15 mg/mL XT-150 | Stage A: 0.45 mg/mL XT-150, Stage B: 0.45 mg/mL XT-150 | Stage A: Placebo, Stage B: 0.15 mg/mL XT-150 | Stage A: Placebo, Stage B: 0.45 mg/mL XT-150
Number analyzed (Participants) | 35 | 35 | 39 | 36 | 36 | 29
score on a scale | -12.73 (2.810) | -12.42 (2.767) | -13.95 (2.695) | -15.28 (2.731) | -9.33 (2.848) | -7.03 (2.904)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent through the last study visit on Day 360 (1 year). Treatment Emergent Adverse Events occurred from the time of study drug treatment on Day 0 through end of study (Day 360) or early termination.
Arm/Group | Stage A: 0.15 mg/mL XT-150, Stage B: 0.15 mg/mL XT-150 | Stage A: 0.15 mg/mL XT-150, Stage B: 0.45 mg/mL XT-150 | Stage A: 0.45 mg/mL XT-150, Stage B: 0.15 mg/mL XT-150 | Stage A: 0.45 mg/mL XT-150, Stage B: 0.45 mg/mL XT-150 | Stage A: Placebo, Stage B: 0.15 mg/mL XT-150 | Stage A: Placebo, Stage B: 0.45 mg/mL XT-150
All-Cause Mortality (participants affected / at risk) | 1/49 | 0/47 | 0/47 | 0/47 | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 3/49 | 2/47 | 3/47 | 2/47 | 4/48 | 3/48
Other Adverse Events (participants affected / at risk) | 15/49 | 16/47 | 18/47 | 24/47 | 10/48 | 23/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage A: 0.15 mg/mL XT-150, Stage B: 0.15 mg/mL XT-150 (N=49) | Stage A: 0.15 mg/mL XT-150, Stage B: 0.45 mg/mL XT-150 (N=47) | Stage A: 0.45 mg/mL XT-150, Stage B: 0.15 mg/mL XT-150 (N=47) | Stage A: 0.45 mg/mL XT-150, Stage B: 0.45 mg/mL XT-150 (N=47) | Stage A: Placebo, Stage B: 0.15 mg/mL XT-150 (N=48) | Stage A: Placebo, Stage B: 0.45 mg/mL XT-150 (N=48)
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage A: 0.15 mg/mL XT-150, Stage B: 0.15 mg/mL XT-150 (N=49) | Stage A: 0.15 mg/mL XT-150, Stage B: 0.45 mg/mL XT-150 (N=47) | Stage A: 0.45 mg/mL XT-150, Stage B: 0.15 mg/mL XT-150 (N=47) | Stage A: 0.45 mg/mL XT-150, Stage B: 0.45 mg/mL XT-150 (N=47) | Stage A: Placebo, Stage B: 0.15 mg/mL XT-150 (N=48) | Stage A: Placebo, Stage B: 0.45 mg/mL XT-150 (N=48)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6) | 7 (8) | 9 (12) | 8 (9) | 3 (3) | 7 (8)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (3) | 2 (2) | 2 (3) | 3 (3) | 2 (3) | 7 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1) | 4 (5) | 0 (0) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 4 (5) | 0 (0) | 3 (4)
Procedural pain (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 3 (3)
COVID-19 (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 5 (5) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 3 (4) | 1 (1) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is bound to terms and conditions of a Sponsored Clinical Trial Agreement which has strict confidentiality obligations running to Sponsor and broad provisions restricting PI's rights to publish or present any data or Study Results without Sponsor's express review consent and review.

DOCUMENTS (2):
  • Study Protocol (2020-03-25): https://cdn.clinicaltrials.gov/large-docs/42/NCT04124042/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-11): https://cdn.clinicaltrials.gov/large-docs/42/NCT04124042/SAP_001.pdf